CLINICAL TRIAL: NCT03928340
Title: Effect of Adding Metformin to Insulin Therapy in Pregnant Women With Type I Diabetes as Regards Pregnancy Outcome
Brief Title: Effect of Adding Metformin to Insulin Therapy on Pregnancy Outcomes in Women With Uncontrolled Type I Diabetes.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Collaborators: Amal Kotb Abdallah (Unknown); Amir Gabr (Unknown); Mohamed Abdeltawwab Mahmoud (Unknown)
Responsible Party: Principal Investigator, Amira S Dieb, Assistant professor, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMBSUREC/05032019/Abd Alaziz
Record Dates: First submitted 2019-04-20; First posted 2019-04-26 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Type1 Diabetes Mellitus
MeSH Terms: interventions — Metformin; Insulin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combined metformin and insulin (Active Comparator)
  Interventions: Drug: Metformin; Drug: Insulin
- Insulin only (Other)
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Metformin — 40 patients will be treated with metformin
  (1 gm twice daily (with the 2 main meals)), combined with insulin therapy
  Arms: combined metformin and insulin
Drug: Insulin — 40 patients will be treated with insulin alone. (Insulin dosage will be adjusted according to endocrinological recommendations)

SUMMARY:
A randomized controlled clinical trial will be conducted in KasrELAiny hospitals, Cairo University and Beni-Suef University Hospital, including 80 uncontrolled diabetic pregnant women (type I) in the 3rd trimester (28-32 weeks of pregnancy) divided equally into study group and control group, to compare the usage of both metformin and insulin instead of using insulin alone. Group assignment will be randomized by computer program.

DETAILED DESCRIPTION:
A total of 80 uncontrolled diabetic pregnant patients in the 3rd trimester seeking medical advice in Beni-Suef University Hospital and meet the eligibility criteria, are approached about participation in the trial and given information pamphlets describing the study. The patients are asked to sign a consent form and will be assigned to one of the 2 groups: Group A (study group); will include 40 patients who will be treated with metformin

(1 gm twice daily (with the 2 main meals)), combined with insulin therapy Group B (control group); will include 40 patients who will be treated with insulin alone. (Insulin dosage will be adjusted according to endocrinological recommendations) All patients will be managed according to NICE guidelines for diabetes with pregnancy (2015) Maternal assessment

* Full history taking Baseline medical history is obtained along with other baseline demographics and concomitant medications including insulin regimen and dose.
* Thorough clinical examination Maternal weight, height and blood pressure measured and recorded.
* Laboratory investigations;

  * Routine labs: CBC, coagulation profile, liver and kidney function at time of participation, 28-32 weeks of gestation especially renal parameter serum Creatinine.
  * HbA1c at time of 1st examination.
  * FBS, 2h post prandial blood sugar will be done weekly from time of participation till time of delivery
* Fundus examination for early detection of retinal affection at Ophthalmology clinic

Follow up:

1. Fetal weight gain weekly
2. Maternal weight gain weekly

Accordingly:

1. Uncontrolled cases will follow up weekly in the High Risk Pregnancy outpatient clinic until 36 weeks and then admitted to High risk pregnancy department for termination of pregnancy

   o Fetal surveillance will be done by ;CTG weekly, Ultrasound weekly and Fetal kick count daily
2. Resistant uncontrolled cases will be admitted to high risk pregnancy department where capillary blood sugar will be measured 7 times daily Fetal surveillance will be done by ; CTG Daily, Ultrasound every 3 days and Fetal kick count daily

Assessment of Patients at time of termination by:

1. Fasting blood sugar , 2 hours post prandial blood sugar and HBA1C
2. Routine preoperative labs. CBC, coagulation profile, liver and kidney function
3. Fetal weight
4. Maternal weight Neonatal assessment after delivery include the following; APGAR score, neonatal weight, incidence of transient tachypnea of newborn (TTN), acute respiratory distress syndrome (ARDS), neonatal hypoglycemia and NICU admission.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic pregnant patients with type one diabetes and no other chronic disorders
* Patients on insulin in the 3rd trimester of pregnancy (on insulin therapy since start of gestation)
* Patients pregnant in single living fetus with no apparent congenital anomalies
* Haemoglobin A 1 C (HbA1c) level between 7% to 11%
* All patients have done a dating ultrasound to confirm gestational age, viability and rule out any abnormality

Exclusion Criteria:

* Patients with type 2 or gestational diabetes
* Patients with intolerance or hypersensitivity to metformin
* Patients with congestive heart failure or a history of congestive heart failure
* Patients with renal insufficiency
* Patients having current significant gastrointestinal problems such as severe vomiting requiring intravenous fluids or hospitalization
* Presence of acute or chronic metabolic acidosis, including diabetic ketoacidosis, a history of diabetic ketoacidosis or history of lactic acidosis
* Patients with liver impairment
* Patients with known higher order pregnancies (twins, triplets, etc.)
* Patients having a known potentially fetal lethal anomaly

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2020-03-29 (Actual); Study Completion 2020-03-29 (Actual)

PRIMARY OUTCOMES:
HbA1c | 12 weeks
  the change in level of glycosylated haemoglobin
capillary glucose | 12 weeks
  the change in level of glucose in capillary blood
fasting blood sugar measurement. | 12 weeks
  the change in level of glucose in venous blood after fasting for 8 hours
2 hours post prandial blood sugar measurement. | 12 weeks
  the change in level of glucose in venous blood 2 hours after meal

SECONDARY OUTCOMES:
Maternal weight gain | 12 weeks
  the change in mothers' weight in kilograms
weekly fetal weight gain measured by ultrasound | 12 weeks
  the change of fetal weight measured by ultrasound
insulin requirements | 12 weeks
  the change in dose of insulin taken by patient
attacks of maternal hypoglycemia | 12 weeks
  Number of patients with plasma glucose level below 65 mg/dl
intra uterine fetal death (IUFD) | 12 weeks
  The number of patients with death of fetus after 20 weeks of gestation
neonatal weight | 12 weeks
  The change in neonatal weight in kilograms
preterm birth | 12 weeks
  The number of patients giving birth berfore 37 completed weeks
neonatal respiratory distress | 12 weeks
  the number of neonates with neonatal respiratory distress
neonatal hypoglycemia | 12 weeks
  the number of neonates with plasma glucose level below less than 45 mg/dL (2.5 mmol/L)
neonatal Intensive care admission | 12 weeks
  the number of neonates with neonatal Intensive care admission

CONTACTS AND LOCATIONS:
Overall Officials: Amal kotb, Principal Investigator — Beniswef university hospital; Amir Gabr, Principal Investigator — Cairo university kasrelainy hospitals
Locations (1):
- Beniswef university hospital, Cairo, Egypt